## PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study

PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study

**Study Unique Protocol ID:** 

3736-1/2022/EKU

**NCT Number:** Not available

## Faculty of Dentistry Department of Oral and Maxillofacial Surgery and Dentistry Director: Dr. habil. PhD Zsolt Németh CONSENT FORM Study Title: PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study Site: Semmelweis University, Department of Oral and Maxillofacial Surgery and Dentistry, 52 Mária St., Budapest, 1085 Principal Investigator: Dr. Martin Major, PhD student, dentoalveolar surgery specialist in training Phone number: daytime phone: +36 70 677 3597 24-hour contact number: +36 1 266 0457 Patient phone number: \_\_\_\_\_ Patient name: \_\_\_\_\_, Date of birth: \_\_\_\_\_ I give my consent to participate in the following clinical study:

## Consent Declaration

The relationship between PRF and BoneAlbumin

SEMMELWEIS UNIVERSITY

I have been satisfactorily informed by my physician, Dr. Martin Major, about the planned surgery, its potential extensions if necessary, and all related information during a detailed consultation. All my questions regarding the surgery, its risks, and possible complications have been answered.

I declare that I fully understand the written and verbal information provided and have no further questions. After sufficient consideration, I consent and request that the offered surgery, with its known and potential risks, be performed on me by the physician.

I will follow the medical instructions required for conducting the clinical trial. However, I understand that my participation is voluntary, and I may withdraw my consent at any time without any adverse effect on my future medical care.

Additionally, I consent to the recording of data collected as part of the clinical study. Representatives of regulatory authorities may review my personal medical records at the hospital to verify the accuracy of the data.

Patient Name in PRINT Date Patient Signature

Responsible Investigator Date Investigator Signature

Name in PRINT

(The patient receives one signed original copy of the Consent Form, and another original copy will be kept in the investigator's site file.)

Address: 52 Mária St., Budapest, 1085

Mailing Address: 26 Üllői Rd., Budapest, 1085; P.O. Box 2, Budapest, 1428

Email: titkarsag.arcallcsont@dent.semmelweis-univ.hu

Phone/Fax: +36 1 266 0456

https://semmelweis.hu/szajsebeszet/